CLINICAL TRIAL: NCT05380492
Title: Phase 1/2a Dose Escalation Study of VOY-101 in Patients With Advanced Non-Neovascular Age-Related Macular Degeneration
Brief Title: Study of VOY-101 in Patients With Advanced Non-Neovascular Age-Related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Perceive Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBI-AMD-001
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Age-related Macular Degeneration; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: The Phase 1 will enroll in a dose escalation study model (three sequential cohorts), followed by a Phase 2a cohort that will be randomized among a maximum tolerated dose arm, a lower dose arm, and a control arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Phase 1 cohorts will be open-label, the Phase 2a cohort will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose (Experimental): VOY-101 Low Dose (single dose, IVT)
  Interventions: Biological: VOY-101
- Mid Dose (Experimental): VOY-101 Mid Dose (single dose, IVT)
  Interventions: Biological: VOY-101
- High Dose (Experimental): VOY-101 High Dose (single dose, IVT)
  Interventions: Biological: VOY-101

INTERVENTIONS:
Biological: VOY-101 — Intravitreal injection of VOY-101

SUMMARY:
This safety study comprises a dose escalation study of VOY-101, followed by a cohort of subjects randomized to the maximum tolerated dose arm, a lower dose arm, and control arm.

DETAILED DESCRIPTION:
This is a prospective, multi-center safety phase 1/2a study to evaluate the safety of a single, unilateral intravitreal (IVT) injection of three dose levels of VOY-101 therapy in subjects with late-stage non-neovascular age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

1. Are ≥50 years of age at the time of consent.
2. Are willing and able to understand and provide written informed consent.
3. Are willing and able to return for scheduled treatment and follow-up examinations.
4. Are able to undergo ETDRS BCDVA testing and ophthalmic imaging.
5. Well-demarcated GA secondary to AMD in the absence of MNV and in the absence of history of MNV.
6. Absence of signs of non-exudative MNV.
7. Additional Ocular Inclusion Criteria
8. Meet certain genotype criteria for risk of AMD.

Exclusion Criteria:

1. Are women of childbearing potential (WOCBP) and are pregnant or unwilling to use and document use of effective contraception for the duration of the study.
2. Additional Systemic, Ocular, and Genetic Exclusion Criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoints | Through 24 months
  1. Frequency of ocular and systemic adverse events (AEs) (serious [SAEs] and treatment-emergent non-serious adverse events [TEAEs])

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Consultants of Texas, Bellaire, Texas
  - University of Utah, Salt Lake City, Utah